CLINICAL TRIAL: NCT00106470
Title: Genetic Epidemiology of COPD in Costa Rica
Brief Title: Genetic Factors That Influence Chronic Obstructive Pulmonary Disease in Hispanics
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1289; R01HL073373 (NIH)
Record Dates: First submitted 2005-03-24; First posted 2005-03-25 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine genetic factors that influence the development of chronic obstructive pulmonary disease (COPD) in Hispanics, a minority group at high risk for the disease.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

This study will concentrate on a genetically isolated Hispanic population with a high prevalence of COPD living in the Central Valley of Costa Rica. Nine hundred individuals from descendants of the Costa Rican Central Valley founder population will be enrolled. To identify regions of the genome that are likely to contain genetic determinants of COPD-related phenotypes in this population, the study will collect phenotypic and genotypic data on 30 large families with a history of moderate to severe COPD that have multiple individuals affected with smoking-related airflow obstruction. A genome scan will be conducted on these individuals using short-tandem repeat (STR) markers. Linkage analysis will be performed on 6 COPD-related phenotypes, which will include the following: 1) chronic bronchitis; 2) airflow obstruction; 3) forced expiratory volume in one second (FEV1); 4) FEV1/FVC[forced vital capacity];5) bronchodilator responsiveness; and 6) total serum immunoglobulin E. Within genomic regions demonstrating linkage to COPD-related phenotypes in the genome scan, narrowly spaced STR markers will be genotyped and tested for linkage between these markers and COPD-related phenotypes. Within selected genomic regions, the association will be tested between single nucleotide polymorphisms (SNPs) in candidate genes and COPD-related phenotypes. By enrolling a large number of participants of a genetically isolated population and utilizing a family-based study design, this study should be able to address an important yet unstudied issue: the genetic influences on the expression of the COPD phenotype in Hispanics.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Reduced FEV1 after administration of bronchodilator (less than or equal to 60% of predicted value)
* At least six great-grandparents born in the Central Valley of Costa Rica
* At least one sibling with a history of smoking (10 or more packs per year)

Exclusion Criteria:

* Chronic respiratory disorder other than COPD (as determined by a questionnaire and high-resolution CT chest scan)
* Severe alpha 1-antitrypsin deficiency

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Families of individuals with physician-diagnosed COPD and smoking-related airflow obstruction who are younger than 71 years.
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2005-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Genetic factors that influence the development of COPD in Hispanics. | Measured through the use of genetic samples

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Celedon, MD, DrPH, Study Chair — University of Pittsburgh
Locations (1):
- Hospital Nacional de Niños, San José, Costa Rica

REFERENCES:
- [Background] Hunninghake GM, Weiss ST, Celedon JC. Asthma in Hispanics. Am J Respir Crit Care Med. 2006 Jan 15;173(2):143-63. doi: 10.1164/rccm.200508-1232SO. Epub 2005 Oct 6. PMID 16210666
- [Background] Brehm JM, Celedon JC. Chronic obstructive pulmonary disease in Hispanics. Am J Respir Crit Care Med. 2008 Mar 1;177(5):473-8. doi: 10.1164/rccm.200708-1274PP. Epub 2007 Nov 20. PMID 18029789
- [Result] Brehm JM, Hagiwara K, Tesfaigzi Y, Bruse S, Mariani TJ, Bhattacharya S, Boutaoui N, Ziniti JP, Soto-Quiros ME, Avila L, Cho MH, Himes B, Litonjua AA, Jacobson F, Bakke P, Gulsvik A, Anderson WH, Lomas DA, Forno E, Datta S, Silverman EK, Celedon JC. Identification of FGF7 as a novel susceptibility locus for chronic obstructive pulmonary disease. Thorax. 2011 Dec;66(12):1085-90. doi: 10.1136/thoraxjnl-2011-200017. Epub 2011 Sep 15. PMID 21921092